CLINICAL TRIAL: NCT03910803
Title: An Open-label Single Center Study to Evaluate the Efficacy of SILIQ™ (Brodalumab) for the Treatment of Moderate Hidradenitis Suppurativa
Brief Title: Treatment of Moderate Hidradenitis Suppurativa
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Florida Academic Dermatology Centers (Other)
Collaborators: Ortho Dermatologics (Industry)
Responsible Party: Principal Investigator, Francisco A. Kerdel, MD, Principal Investigator, Florida Academic Dermatology Centers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2018-3620
Record Dates: First submitted 2019-03-29; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brodalumab - Open Label (Other): Randomized subjects will be receiving Brodalumab (210 mg) administered by subcutaneous injection at the following visits: Baseline, week 1, week 2 and every two weeks thereafter, until Week 24.
  Investigational Product not to be administer into areas where the skin is tender, bruised, red, hard, thick, scaly, or affected by Hidradenitis Suppurativa.
  Interventions: Drug: Brodalumab

INTERVENTIONS:
Drug: Brodalumab — Brodalumab is a human monoclonal IgG2κ antibody directed against human interleukin-17 receptor A (IL-17RA). It is expressed in a Chinese Hamster Ovary (CHO) cell line. Brodalumab is comprised of 1312 amino acids and has an estimated molecular mass of 144,000 Daltons.
  Brodalumab Injection is a sterile, preservative-free, yellow solution, delivered via subcutaneous injection. . Each Brodalumab single dose prefilled syringe delivers 1.5 mL of solution containing 210 mg of brodalumab formulated in glutamate (6.5 mg), polysorbate 20 (0.15 mg), proline (36 mg), and Water for Injection, USP at pH 4.8.
  Other Names: Siliq

SUMMARY:
The study will be conducted over 24 weeks on active therapy followed by a four-week observational visit. The total length of the study will be 28 weeks.

Study visits will occur at Screening, Baseline (Week 0), Weeks 4, 8, 12, 16, 20, 24 followed by an observational visit. Additionally, all subjects will be contacted by phone 1 week following the Baseline visit to ensure daily pain assessments are being recorded. If any signs or symptoms are reported at the time of the call, an unscheduled study visit will be conducted to assess whether an infection is present.

Adverse events will be collected throughout the study.

DETAILED DESCRIPTION:
An Open-label Single Center Study to Evaluate the Efficacy of SILIQ™ (brodalumab) for the Treatment of Moderate Hidradenitis Suppurativa. In this Single-Center study a total of 20 subjects will be randomized for a period of 24 weeks of treatment, Followed by an observational four-week post treatment visit. Study visits will occur at Screening , Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 28 (4 weeks off therapy). Additionally, all subjects will be contacted by phone 1 week following the Baseline visit to ensure daily pain assessments are being recorded. If any signs or symptoms are reported at the time of the call, an unscheduled study visit will be conducted to assess whether an infection is present.

At Week 4 or Week 8, if PGA is greater or equal to 2 points of baseline, antibiotic rescue is permitted (minocycline or doxycycline up to 100 mg bid).

Safety and efficacy measurements will be performed throughout the study.

The duration of the screening period will be a minimum of 7 days and a maximum of 30 days during which time all of the inclusion and exclusion criteria will be evaluated.

Subjects will have up to 30 days to return to the site for the Baseline visit from the date of the Screening visit.

No study drug will be administered at the final visit.

Subjects may discontinue treatment at any time during study participation. Subjects who prematurely discontinue will be asked to complete a early termination visit.

Subjects who initially screen fail for the study may be permitted to re-screen following re-consent. All screening procedures with the possible exceptions noted below will be repeated. The subject must meet all inclusion and none of the exclusion criteria at the time of re-screening in order to qualify for the study.

The protocol of the study will be approved by the Institutional Review Board (IRB) or the Ethics Committee (EC) of the participating study sites. Depending on the participating countries both local and central IRB/EC approvals will be granted. The study will be registered at www.clinicaltrials.gov before the enrollment of the first patient. The trial will be conducted in compliance with the protocol, GCP, and all applicable regulatory requirements.

Study Endpoints

Primary Endpoint:

The Proportion of subjects achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at week 16, defined as a 50% reduction in the total number of abscess and inflammatory nodule count as long as the fistulae and abcess count remains the same.

Secondary Endpoints:

* The number of patients achieving a one point reduction in PGA score at week 16
* Changes in Modified Sartorius scale from Baseline to Week 16
* The number of patients achieving a two point reduction (required from baseline score) in VAS pain score at week 16
* Dermatology Life Quality Index or DLQI,

ELIGIBILITY:
Inclusion Criteria:Subjects are included in the study if they meet all of the following criteria:

* Written informed consent provided by the patient.
* Male or female, at least 18 years of age..
* Subject must be in general good health ( except for Hidradenitis Suppurativa) as judged by the Investigator, based on medical history, physical examination, clinical laboratories and urinalysis. NOTE: the definition of good health means a subjects that does not have uncontrolled significant co-morbid conditions.
* Must have a diagnosis of HS for at least 6 months prior to Baseline/Screening visit
* Subjects with moderate HS with a PGA score of 3 defined as having: 0 abscesses, 0 draining fistula, and 5 inflammatory nodules; or 1 abscess or draining fistula and 1 inflammatory nodule; or 2-5 abscesses or draining fistulas and 10 inflammatory nodules
* HS lesions must be present in at least two distinct anatomic areas, one of which must be at least Hurley Stage II (see definition of terms)
* Subject must have stable HS for at least 2 months (60 days) prior to Screening/ Baseline visit as determined by the investigator through subject interview and review of medical history;
* Subject must have a total abscess and inflammatory nodule (AN) count (PGA) of no greater than moderate at the Baseline visit. Patient with PGA 0-1 (No disease or minimal Disease will be excluded).
* Subject must agree to daily use (and throughout the entirety of the study) of one of the following over-the-counter topical antiseptics on their HS lesions: chlorhexidine gluconate, triclosan, benzoyl peroxide, or dilute bleach in bathwater.
* Women who are postmenopausal must have a negative serum pregnancy test on entry in the study.
* Females of childbearing potential (FCBP)† must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive§ options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).

The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).

* The screening/baseline laboratory test results must meet the following criteria (WNL means within normal limits for patients with HS [e.g., may have slightly higher WBC and platelet counts]):
* WBC (white blood cell count): WNL
* ANC (absolute neutrophil count): WNL
* Hemoglobin: >10 mg/dl
* Platelets: WNL
* Serum Creatinine: WNL
* SGOT (AST - aspartate aminotransferase): <2 times upper normal limit
* SGPT (ALT - alanine aminotransferase): <2 times upper normal limit
* Alkaline phosphatase:<2 times upper normal limit

Exclusion Criteria:

Subjects with ANY of the following will be excluded from the study:

* The presence of any of the following will exclude a subject from enrollment:
* Subjects with PGA 4 and 5 , with 15 lesions and significant scarring (defined as any linear, indurated area, extended across more than 50% of the circumference of the affected area) ,fistulas or sinus tract involvement will be excluded.
* Other than Hidradenitis Suppurativa , any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
* Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last study drug dose (this includes father's who plan on fathering a child within 6 months after their last study drug dose.
* Active substance abuse or a history of substance abuse within 6 months prior to Screening
* Malignancy or history of malignancy, except for: treated [ie, cured] basal cell or squamous cell in situ skin carcinomas; treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
* Active substance abuse or a history of substance abuse within 6 months prior to Screening. .
* Patient with diagnosis or suspected Crohns disease or Ulcerative Colitis.
* Patient who is on a stable dose of analgesics, will be allowed to remain on them. No new opiates will be permitted during the trial.
* Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
* Prior treatment with Anti IL-17 drugs ( Secukinumab, ixekizumab and Brodalumab)
* Known allergy to Brodalumab
* Have a known history of serious infections (eg, hepatitis, pneumonia or pyelonephritis) in the previous 3 months
* Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (eg, nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access
* Patient with significant scarring, fistulas, or sinus tract involvement will be excluded. Only subjects with inflammatory abscesses and nodules will be allowed to enter the study.
* Infection(s) requiring treatment with intravenous (IV) anti-infectives (antibiotics, antivirals, antifungals) within 30 days prior to Baseline or oral anti-infectives (antibiotics, antivirals, antifungals) within 14 days prior to Baseline
* Any other active skin disease or condition (e.g., bacterial, fungal or viral infection) that may interfere with assessment of HS;
* History of invasive infection (e.g., listeriosis, histoplasmosis), human immunodeficiency virus (HIV);
* Subject has an active systemic viral infection or any active viral infection that based on the investigator's clinical assessment make the subject an unsuitable candidate for the study;
* Hepatitis B: HBsAg positive (+) or detected sensitivity on the HBV-DNA PCR qualitative test for HBc Ab/HBsAb positive subjects; Or Hepatitis C
* Chronic recurring infections or active TB;
* Evidence of dysplasia
* Pregnant (or considering becoming pregnant) or lactating females.
* The use of any prior biologic therapy is prohibited
* Subjects currently undergoing any of the following treatments for HS will require a 2 week wash-out period: Minocycline; Tetracycline; Clindamycin; Rifampicin and Steroids.
* Presence of active suicidal ideation, or positive suicide behavior using Columbia Suicide Severity Rating Scale (eC-SSRS) and with either of the following criteria: History of a suicide attempt within the 5 years prior to the Screening Visit; Subjects with a history of a suicide attempt more than 5 years ago should be evaluated by a mental healthcare practitioner (HCP) before enrolling into the study. Suicidal ideation in the past month prior to the Screening Visit as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the of the C-SSRS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response (HiSCR) | Study assessments occurr at baseline and at weeks 4, 8, 12, 16, 20, 24, and 28"
  Patients at week 16 achieving the Hidradenitis Suppurativa Clinical Response (HiSCR), defined as a ≥ 30% reduction in the total number of abscess and inflammatory nodules, with no increase in the number of abscesses or draining fistulas.
Hidradenitis Suppurativa Clinical Response (HiSCR30) | Study assessments occurr at baseline and at weeks 4, 8, 12, 16, 20, 24, and 28"
  Patients at week 16 achieving the Hidradenitis Suppurativa Clinical Response (HiSCR), defined as a ≥ 30% reduction in the total number of abscess and inflammatory nodules, with no increase in the number of abscesses or draining fistulas. (HiSCR30) when compared with baseline.
Hidradenitis Suppurativa Clinical Response (HiSCR50) | Study assessments occurr at baseline and at weeks 4, 8, 12, 16, 20, 24, and 28"
  Patients achieving a ≥ 30% and ≥ 50% reduction in HiSCR at week 24;

SECONDARY OUTCOMES:
Physician s Global Assessment ( PGA) | Study assessments occurr at baseline and at weeks 4, 8, 12, 16, 20, 24, and 28"
  The PGA score is based on a cumulative global assessment of nodule, abscess, and fistula counts corresponding to a 5-point score (0 = clear, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe). Efficacy endpoint : the proportions of patients achieving a 1-point reduction in the PGA score.
Modified Sartorius | Study assessments occurr at baseline and at weeks 4, 8, 12, 16, 20, 24, and 28"
  The modified Sartorius score consists of 4 clinical parameters including the number of affected areas and HS lesion hallmarks. It has a minimum value of 0 and no maximum limit.8 Efficacy endpoint :Changes in Modified Sartorius scale from Baseline to Week 16
VAS | Study assessments occurr at baseline and at weeks 4, 8, 12, 16, 20, 24, and 28"
  Pain will be assessed using a 100-mm VAS (0 = no pain, 100 = maximum pain). The number of patients achieving a two point reduction (required from baseline score) in VAS pain score at week 16
Dermatology Life Quality Index or DLQI | Study assessments occurr at baseline and at weeks 4, 8, 12, 16, 20, 24, and 28"
  It is a validated and widely used questionnaire for assessing Quality of Life related to dermatology conditions. Its score constitutes the summation of responses to all 10 items, ranging from 0 (the best QoL) to 30 (worse QoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Academic Centers Research and Education, LLC, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No